CLINICAL TRIAL: NCT02187653
Title: Spine Registry Exposure for: Lumbar and Cervical Surgery Utilizing IOM
Brief Title: Intraoperative Monitoring (IOM) Patient Registry
Acronym: IOM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: DC2 Healthcare (Industry)
Collaborators: National Neurosurgical and Orthopedic Optimum Care Continuum (NOC2) Foundation (Unknown); National Research Independent Operations Management (Other)
Responsible Party: Sponsor
Other Study IDs: DOC 1002
Record Dates: First submitted 2014-07-07; First posted 2014-07-11 (Estimated); Last update posted 2014-07-11 (Estimated); Status verified 2014-07

CONDITIONS: Intraoperative Monitoring; Spinal Diseases
Keywords: IOM; IONM; Intraoperative Monitoring; Intraoperative Neuromonitoring; Spine; Lumbar; Cervical
MeSH Terms: conditions — Spinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lumbar: Patients undergoing lumbar surgery
- Cervical: Patients undergoing cervical surgery

SUMMARY:
The primary objective of this study is to evaluate the rate of new or worsening neurologic deficits and/or radiculopathy following lumbar or cervical surgery in light of IOM using neurological testing (motor and sensory) in the optimal management of the surgical patient.

DETAILED DESCRIPTION:
Prospective reports will be collected on approximately 10,000 patients undergoing lumbar or cervical spinal surgery using intraoperative monitoring. Patients will be enrolled in registry after signing informed consent. Data will be collected prior to surgery, during surgery, immediately following surgery and 4 to 6 weeks post surgery. The registry will serve as a database for surgeries using IOM.

Specific outcome measures will be: neurological assessment, length of hospital stay, pain intensity, and complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar or cervical surgery
* Utilization of IOM
* Understand and sign informed consent

Exclusion Criteria:

* There are no specific exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cervical or lumbar surgery in which intraoperative monitoring has been utilized.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2011-09; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Neurological Assessment at 24 hours | baseline and 24 hours from time of surgery
  Motor, Reflex, and Sensory testing will be assessed for change from baseline and 24 hours after surgery
Change in Pain Intensity from Baseline at 24 hours | baseline and 24 hours from time of surgery
  Pain intensity will be measured by Visual Analogue Scale (VAS) for change from baseline and 24 hours after surgery
Complications | At time of surgery
Change from baseline in Neurological Assessment at 6 weeks | baseline and 6 weeks
  Motor, Reflex, and Sensory testing will be assessed for change from baseline, within 6 weeks but not less than 4 weeks
Change in Pain Intensity from Baseline at 6 weeks | baseline and 6 weeks
  Pain intensity will be measured by Visual Analogue Scale (VAS) within 6 weeks but not less than 4 weeks
Complications | 24 hours after surgery
Complications | 6 weeks after surgery
  within 6 weeks after surgery but not less than 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- DC2 Healthcare, Nashville, Tennessee, United States

REFERENCES:
- See also: DC2 Healthcare — http://www.dc2healthcare.com
- See also: NRIOM — http://www.nriom.com/